CLINICAL TRIAL: NCT07028580
Title: Evaluation of a High Protein Plant Dominant Diet (HiProPlaDo) in Sarcopenia, Quality of Life and Metabolic Parameters in Patients With Liver Cirrhosis: A Randomized Clinical Trial
Brief Title: Evaluation of a High Protein Plant Dominant Diet (HiProPlaDo) in Liver Cirrhosis
Acronym: HiProPlado
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Kalliopi Anna Poulia, Assistant Professor in Clinical Dietetics, Agricultural University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 227 15/4/2022
Record Dates: First submitted 2025-03-21; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-03

CONDITIONS: Liver Diseases; Cirrhosis, Liver; Sarcopenia; Malnutrition; Cachexia
Keywords: malnutrition; plant based diet; protein; sarcopenia; liver disease
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis; Sarcopenia; Malnutrition; Cachexia

STUDY DESIGN:
Intervention Model Description: Double Blind randomized clinical trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (diet with animal protein). (Experimental): In group Α, a diet was designed based on the needs of each individual, based on proteins of animal origin.
  Interventions: Other: Diet based on animal proteins
- Group B (diet with plant based protein). (Experimental): In group B, a diet was designed based on the needs of each individual, based on proteins of plant origin.
  Interventions: Other: Diet based on plant proteins.
- Group C (control) (Other): Control group who were given general instructions for patients with liver disease.
  Interventions: Other: General instructions for patients with liver disease.

INTERVENTIONS:
Other: Diet based on animal proteins — Ιntervention with a diet based on animal proteins.
  Arms: Group A (diet with animal protein).
Other: Diet based on plant proteins. — Ιntervention with a diet based on animal proteins.
  Arms: Group B (diet with plant based protein).
Other: General instructions for patients with liver disease. — Α brochure with general instructions was designed for patients with liver disease.
  Arms: Group C (control)

SUMMARY:
The aim of the study is to compare the implementation of a high-protein diet based on plant-based foods (Group A) with the usual guidelines for liver patients, in which protein needs are met by low-fat animal foods (Group B). The parameters that will be studied concern:

1. Liver function
2. Nutritional status and the risk of malnutrition
3. Body composition, with emphasis on muscle mass

3. Muscular system functionality and sarcopenia 4. The intestinal microbiome 5. The quality of life of the patients

This is a randomized, double-blind intervention study lasting 6 months, during which volunteers will be asked to answer, with the help of the researchers, questionnaires assessing nutritional risk, assessing physical activity and quality of life, and assessing nutritional intake (24-hour food recall and Food Frequency Questionnaire). At the same time, a blood sample will be collected for analysis of inflammatory factors and indicators related to nutritional status (albumin, prealbumin, cholesterol, total iron binding capacity). Body composition will be assessed using the method of anthropometry and dual-energy X-ray absorptiometry (DEXA), and hand dynamometry to assess functionality. The assessment of the microbiome will be performed by saliva collection and/or stool collection. The impact on liver function will be assessed by recording every 3 months a) natriuresis/microalbuminuria (in 24-hour urine collection or urine sample) and the severity of ascites (grade I, II, III), b)ammonia levels and episodes of encephalopathy, c) complications of cirrhosis, such as variceal hemorrhage, encephalopathy, spontaneous bacterial peritonitis and renal dysfunction, d) liver disease severity assessment scores, such as MELD and Child-Pugh scores.

The aim of the study is to see if there is a difference in sarcopenia and the values of various biochemical indicators between patients who received plant-based proteins compared to patients who received animal-based proteins.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with decompensated cirrhosis awaiting kidney transplantation who have not previously received dietary advice.

Exclusion Criteria:

* Psychopathological illness
* Adoption of a vegetarian diet prior to study entry
* Hepatonephrotic syndrome requiring protein restriction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measurements | From the first day and 3 months later
  The following parameters will be measured and combined into various equations to evaluate the body weight and body composition of each patient, body weight (kg) , height (m^2) , mid-arm circumference (cm) , skinfolds (mm), dynamometry and biochemical/hematological testing were performed.
Quality of life (QoL) assessment | From the first day and 3 months later
  Quality of life (QoL) was assessed with the SF-36 questionnaire.
Dietary compliance | From the first day and 3 months later
  Dietary compliance was assessed with 24-hour recalls and a food frequency questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Laikon General Hospital of Athens, Athens, Attica
  - Agricultural University of Athens, Athens, Attica

IPD SHARING:
Plan to Share IPD: Yes